CLINICAL TRIAL: NCT02126267
Title: Clinical and Microbiological Evaluation of Techniques for Scaling and Root Planing Per Quadrant and One Stage Full Mouth Disinfection Associated With Azithromycin or Chlorhexidine: Randomized Controlled Trial
Brief Title: Evaluation of Techniques for Scaling and Root Planing and One Stage Full Mouth Disinfection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Lavras (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Douglas Campideli Fonseca, Master of Science, Centro Universitario de Lavras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07172212.3.0000.5149
Record Dates: First submitted 2014-04-21; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Periodontal Disease; Chronic Periodontitis
Keywords: periodontal disease; therapy; anti-bacterial agents; Randomized Controlled Trials
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; gluconic acid; Azithromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Full mouth disinfection - FMD (Experimental): n = 10: Procedures for scaling and root planing were performed in a single stage (24 hours) divided into two sessions (60 min per session) on two consecutive days
  Interventions: Procedure: Full mouth disinfection
- FMD + chlorhexidine (FMD-CX) (Experimental): n = 15: Same as FMD with the inclusion of chlorhexidine in office (application of chlorhexidine (CX) (1%) gel in pockets after scaling, brushing tongue for 1 min. with CX (1%) gel and mouthwash at the beginning and end of each session with CX 0.2% for 30 seconds (with the form of a gargle in the last 10 seconds)). In addition, use was made of homemade CX 0.2% for 60 days after the scaling in a single phase.
  Interventions: Procedure: Full mouth disinfection; Drug: Chlorhexidine gel and gluconate; Drug: Chlorhexidine gluconate solution
- FMD + azithromycin (FMD-AZ) (Experimental): n = 15: Same as with the FMD include the use of azithromycin (500 mg) once daily for 3 consecutive days. Medication was started the same day as the end of the scaling.
  Interventions: Procedure: Full mouth disinfection; Drug: Azithromycin
- Scaling and root planing (SRP) (Experimental): (n = 13): scaling procedures were performed per quadrant (30 min. per quadrant) at weekly intervals between sessions;
  Interventions: Procedure: Scaling and root planing
- SRP + azithromycin (SRP-AZ) (Experimental): n = 11: Same as scaling and root planing group (SRP) with inclusion of the use of azithromycin (500 mg) once daily for 3 consecutive days. Medication was started the same day as the end of the last scaling hemi-arch;
  Interventions: Procedure: Scaling and root planing; Drug: Azithromycin
- SRP + chlorhexidine (SRP-CX) (Experimental): n = 13 : Same as group scaling and root planing (SRP) with the inclusion of home use of CX 0.2% for 60 consecutive days after the end of the first session of scaling
  Interventions: Procedure: Scaling and root planing; Drug: Chlorhexidine gluconate solution

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling procedures were performed per quadrant (30 min. per quadrant) at weekly intervals between sessions;
  Arms: SRP + azithromycin (SRP-AZ); SRP + chlorhexidine (SRP-CX); Scaling and root planing (SRP)
Procedure: Full mouth disinfection — Procedures for scaling and root planing were performed in a single stage (24 hours) divided into two sessions (60 min per session) on two consecutive days
  Arms: FMD + azithromycin (FMD-AZ); FMD + chlorhexidine (FMD-CX); Full mouth disinfection - FMD
Drug: Chlorhexidine gel and gluconate — application of chlorhexidine (CX) (1%) gel in pockets after scaling, brushing tongue for 1 min. with CX (1%) gel and mouthwash at the beginning and end of each session with CX 0.2% for 30 seconds (with the form of a gargle in the last 10 seconds)
  Arms: FMD + chlorhexidine (FMD-CX)
Drug: Chlorhexidine gluconate solution — Home use fo CX 0.2% for 60 consecutive days after the end of the first session of scaling.
  Arms: FMD + chlorhexidine (FMD-CX); SRP + chlorhexidine (SRP-CX)
Drug: Azithromycin — Azithromycin (500 mg) once daily for 3 consecutive days.
  Arms: FMD + azithromycin (FMD-AZ); SRP + azithromycin (SRP-AZ)

SUMMARY:
Evaluate and compare the effectiveness in a clinical and microbial perspective one stage full-mouth disinfection technique in relation to scaling and root planing per quadrant associated with chlorhexidine or azithromycin.

DETAILED DESCRIPTION:
Seventy -seven systemically healthy subjects with chronic periodontitis were randomly included in 6 different predefined groups. The following periodontal parameters were evaluated: probing depth , clinical attachment level , plaque index, gingival index and percentage of areas affected by periodontal disease. Microbiologically were evaluated the bacterial load and specific load of five bacterias: The quantification of the bacteria was performed by real-time Polymerase Chain Reaction . The clinical and microbial baseline evaluations were performed ( periodontal pre- therapy) , 90 and 180 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of slight-moderate chronic periodontitis

Exclusion Criteria:

* Those who were making regular use of antibiotics or anti-inflammatory drugs or had done up to three months before the beginning of the study;
* those who were making regular use (twice a day) of oral rinses with chlorhexidine or essential oils or have made regular use within three months prior to study entry;
* individuals with a history of sensitivity to chlorhexidine or azithromycin;
* subjects undergoing periodontal therapy include dental scaling procedures in the 12 months preceding the start of the study;
* subjects with impaired bifurcation or trifurcation class III;
* who required antibiotic prophylaxis for conducting clinical periodontal examination
* subjects with removable partial dentures and removable or fixed orthodontic appliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in clinical attachment | Baseline and 180 days after treatment
  In this parameter we will evaluate the distance from the cement-enamel junction to the bottom of the periodontal pocket or gingival sulcus. This measurement is made with a periodontal probe graduated in millimeters

SECONDARY OUTCOMES:
Change in probing depth | Baseline and 180 days after treatment
  In this parameter we will evaluate the distance between the gingival margin and the bottom of the periodontal pocket or gingival sulcus. This measurement is made with a periodontal probe graduated in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Fonseca, Ms, Principal Investigator — Universitary Center of Lavras
Locations (1):
- Douglas Campideli Fonseca, Lavras, Minas Gerais, Brazil

REFERENCES:
- [Result] Emingil G, Han B, Ozdemir G, Tervahartiala T, Vural C, Atilla G, Baylas H, Sorsa T. Effect of azithromycin, as an adjunct to nonsurgical periodontal treatment, on microbiological parameters and gingival crevicular fluid biomarkers in generalized aggressive periodontitis. J Periodontal Res. 2012 Dec;47(6):729-39. doi: 10.1111/j.1600-0765.2012.01488.x. Epub 2012 May 9. PMID 22571226